CLINICAL TRIAL: NCT04970342
Title: Validation of the Drug Impaired Driving Scenario (DIDS) on the CRCDS-miniSim: Evaluating Sensitivity to the Effects of Cannabis and Alprazolam
Brief Title: Validation of the Drug Impaired Driving Scenario (DIDS) on the CRCDS-miniSim
Acronym: PDID
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Timothy L. Brown (Other)
Collaborators: National Highway Traffic Safety Administration (NHTSA) (U.S. Federal Agency); Acclaro Research Solutions, Inc. (Industry); Cognitive Research Corporation (Industry)
Responsible Party: Sponsor-Investigator, Timothy L. Brown, Director of Drugged Driving Research, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 202105389
Record Dates: First submitted 2021-06-24; First posted 2021-07-21 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2022-08

CONDITIONS: Driving Behavior; Driving Under the Influence
Keywords: Driving; Cannabis; Xanax; Marijuana; Alprazolam; Driving Impairment; Substance Use; SDLP; CogScreen; CRCDS
MeSH Terms: conditions — Driving Under the Influence; Marijuana Abuse; Substance-Related Disorders | interventions — Lactose; Capsules; Alprazolam; nabiximols; Dronabinol

STUDY DESIGN:
Intervention Model Description: The study uses two treatments - alprazolam and cannabis - and placebo. Subjects are randomized to a study sequence where the order of treatments (study arm) is counter-balanced, but all treatments and placebo are received by all subjects. At a visit, you might receive placebo alprazolam and placebo cannabis, placebo alprazolam and active cannabis, or active alprazolam and placebo cannabis. There is not a visit where you receive both active alprazolam and active cannabis.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study Site/National Advanced Driving Simulator: Triple (Participant, Investigator, Outcomes Assessor) blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- "Sober" or Double Placebo (Experimental): Subject receives alprazolam capsule containing placebo (lactose). Subject receives placebo cannabis (0% THC / 0% CBD).
  Interventions: Drug: Placebo (Lactose) Capsule; Drug: Cannabis (0%/ THC / 0% CBD)
- Active Alprazolam (Xanax), Placebo Cannabis (Experimental): Subject receives active 0.75 mg alprazolam capsule. Subject receives placebo cannabis (0% THC / 0% CBD).
  Interventions: Drug: 0.75 mg Alprazolam Capsule; Drug: Cannabis (0%/ THC / 0% CBD)
- Placebo Alprazolam (Xanax), Active Cannabis (Experimental): Subject receives alprazolam capsule containing placebo (lactose). Subject receives active cannabis (6.18% THC / <0.025% CBD).
  Interventions: Drug: Placebo (Lactose) Capsule; Drug: Cannabis (6.18% THC / <0.025% CBD)

INTERVENTIONS:
Drug: Placebo (Lactose) Capsule — Single dose on two of the three study visits, orally administered 40 minutes prior to cannabis dose
  Other Names: Placebo; Placebo Alprazolam
  Arms: "Sober" or Double Placebo; Placebo Alprazolam (Xanax), Active Cannabis
Drug: 0.75 mg Alprazolam Capsule — Single dose on one of the three study visits, orally administered 40 minutes prior to cannabis dose
  Other Names: Xanax; Active Alprazolam; Active Xanax
  Arms: Active Alprazolam (Xanax), Placebo Cannabis
Drug: Cannabis (6.18% THC / <0.025% CBD) — Cannabis vapor is produced from 500 mg of dried plant material (6.18% THC / <0.025% CBD). Subjects will inhale using the Foltin Puff Procedure over 10 minutes. Single inflated bag/dose consumed via inhalation 40 minutes after alprazolam dose on one of the three study visits.
  Other Names: Marijuana; Marihuana; Active Cannabis
  Arms: Placebo Alprazolam (Xanax), Active Cannabis
Drug: Cannabis (0%/ THC / 0% CBD) — Cannabis vapor is produced from 500 mg of dried plant material (0% THC / 0% CBD). Subjects will inhale using the Foltin Puff Procedure over 10 minutes. Single inflated bag/dose consumed via inhalation 40 minutes after alprazolam dose at two of the three study visits.
  Other Names: Marijuana; Marihuana; Placebo Cannabis; Placebo
  Arms: "Sober" or Double Placebo; Active Alprazolam (Xanax), Placebo Cannabis

SUMMARY:
Subjects will participate in a 4-visit study protocol at the National Advanced Driving Simulator, part of the University of Iowa, in which they will be asked to complete assorted questionnaires, computerized cognitive tasks, and a simulator drive. Subjects will be administered 0.75 mg alprazolam (Xanax) or placebo and 500 mg vaporized cannabis (6.18% THC / <0.025% CBD) or placebo (0% THC / 0% CBD).

The primary objective of this study is to validate the Drug Impaired Driving Scenario (DIDS) using the CRCDS-2 driving simulator by assessing the acute effects of cannabis relative to placebo on simulated driving performance. Assay sensitivity will be demonstrated by the significant effect of 0.75 mg alprazolam (active comparator) on driving and cognitive endpoints.

DETAILED DESCRIPTION:
At the University of Iowa's National Advanced Driving Simulator (NADS), normal healthy subjects who currently use cannabis recreationally (at least once a month) will be recruited. The study involves four visits, the first of which is a screening visit of approximately 3 hours. At the screening visit, consent is obtained, questionnaires are given, and a physical and psychological exam is administered. Subjects will also train on study procedures, such as the cognitive testing, the simulator drive, and the cannabis inhalation procedure. Subjects will then be scheduled for their three treatment visits, which will be one week apart..

The treatment visits will have a clean (double placebo) and two treatment visits (active alprazolam and placebo cannabis, placebo alprazolam and active cannabis). The alprazolam dose is 0.75 mg and the cannabis dose is 500 mg. All cannabis will be inhaled via a Volcano® Digit vaporizer using the Foltin Puff Procedure. Each of the treatment visits will last approximately twenty-three hours and will include intake with eligibility and baseline testing, transport to a local hotel, an overnight stay at the hotel, transport to NADS, being dosed with study drugs or placebos, cognitive assessments, a simulator drive, and assorted questionnaires. There will also be 8 mL blood sampling before dosing, before driving, and after driving. Each randomized subject will complete a treatment visit of each type one week apart in a counterbalanced sequence.

Meals will be provided at the treatment visits (dinner, snack, breakfast, lunch). Subjects will be monitored until the drug effects have subsided sufficiently to ensure it is safe to transport them home. Subjects will need to arrange their own transportation; they will not be permitted to drive themselves home after the treatment visits.

ELIGIBILITY:
Inclusion Criteria:

* Understands and provides written informed consent prior to the initiation of any protocol-specific procedures.
* Able to comprehend and willing to comply with the requirements of the protocol.
* Healthy male or female adult, 19 to 45 years of age, inclusive, at Screening.
* Regular sleep pattern (usual bedtime between 21:00 and 00:00).
* Score <10 on Epworth Sleepiness Scale at Screening.
* Able to reliably perform study assessments at Screening (On practice scenario, SDLP no higher than 1 standard deviation greater than the mean for normal healthy adults completing the practice scenario and subject has 7 or more correct hits on the Divided Attention task; CogScreen SDC Correct no less than 1 standard deviation below the mean for healthy adults); demonstrates the ability to understand task instructions at Screening; and is physically (e.g., adequate manual dexterity, vision, and hearing) and cognitively capable of performing study tasks at Screening.
* Possesses (and is willing to provide) a valid driver's license and is an active driver.
* Determined to be (by self-report) an active cannabis user with use of at least once per month over the preceding 90 days.
* Willing to abstain from cannabis use (other than study drug) beginning at the end of Screening until discharge from NADS on Day 2 of Treatment Period 3.
* Female subjects must meet one of the following criteria: 1) If of childbearing potential, female subjects agree to use two contraceptive regimens or remain abstinent during the study; or 2) if of non-childbearing potential, female subjects should be surgically sterile or in a menopausal state.

Exclusion Criteria:

* A significant history and/or presence of hepatic, renal, cardiovascular, pulmonary, neurological, psychiatric, gastrointestinal, hematological, immunologic, ophthalmologic, metabolic, or oncological disease, or any other medical issue that would, in the opinion of the Investigator, present undue risk for the subject in the study.
* A history of suicidal behavior within 24 months of Screening, has answered YES to questions 3, 4, or 5 on the C-SSRS at Screening or at any clinic admission, or is currently at risk of suicide in the opinion of an Investigator.
* A recent history (within 6 months prior to Screening) of substance use disorder (including alcohol) (as judged by the Investigator) or regularly consumes >2 alcoholic drinks/day during the last 3 months prior to Screening (1 alcoholic drink is approximately equivalent to: beer [284 mL], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]). Subjects who consume 3 drinks per day but less than 14 drinks per week may be enrolled at the discretion of the Investigator.
* Demonstrates simulator sickness questionnaire scores which are indicative of simulator sickness as defined in the driving simulation operations manual.
* Regularly consumes excessive amounts of caffeine, defined as greater than 6 servings of coffee, tea, cola, or other caffeinated beverages per day.
* Smokes more than 10 cigarettes or e-cigarettes, or 3 cigars or pipes per day, or is unable to refrain from smoking during study visits.
* Has been exposed to an investigational drug or device within the 30 days, or 5 half lives (if known), whichever is longer, prior to Screening.
* Has used a prescription or over-the-counter medication known to cause sedation within 7 days prior to Admission for Period 1 and is unwilling or unable to refrain from sedating medication use during study participation.
* Has used any benzodiazepine, barbiturate, or GABAA modulator (e.g., eszopiclone, zopiclone, zaleplon, and zolpidem) within 28 days prior to Admission for Period 1 or is unwilling or unable to refrain from medication use during study participation.
* Has a history of hepatitis B surface antigen, hepatitis C antibodies, or human immunodeficiency virus (HIV) antibodies 1 or 2.
* Is pregnant or breastfeeding at Screening or any clinic admission or will attempt to become pregnant at any time during study participation.
* Has a clinically significant abnormal finding on 6-lead electrocardiogram (ECG) at Screening or at any clinic admission. The ECG may be repeated once for confirmatory purposes if initial values obtained exceed the limits specified.
* Has a positive urine test for drugs of abuse (other than tetrahydrocannabinol (THC)) or Breath Alcohol Concentration (BrAC) > 0.0 at Screening or any admission.
* Has any clinically significant abnormal physical examination finding at Screening or any clinic admission.
* Participates in night shift work.
* Has traveled across ≥1 time zone in the 2 weeks prior to Admission for Period 1 or is expected to travel across ≥1 time zone during the study.
* Is investigative site personnel or their immediate families (spouse, parent, child, or sibling whether biological or legally adopted).

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2021-08-21 (Actual); Study Completion 2021-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L Brown, Principal Investigator — National Advanced Driving Simulator, University of Iowa
Locations (1):
- National Advanced Driving Simulator, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
Data is being collected to support regulatory efforts by the government and data will not be available to those outside of the research team and government at this time.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 13 subjects enrolled, 8 were randomized to one of six sequences counterbalancing the three treatment arms. Subjects were randomized at intake for Treatment Visit 1. Of the 5 subjects enrolled but not randomized, 3 did not meet study criteria at the screening visit, 1 had scheduling conflicts, and 1 failed to show for Treatment Visit 1. There was a minimum 7-day washout between the Screening Visit and intake for Treatment Visit 1. All randomized subjects completed all treatment arms.
Groups:
- Sequence 1: Treatment Visit 1: Experimental: "Sober" or Double Placebo Subject receives alprazolam capsule containing placebo (lactose). Subject receives placebo cannabis (0% THC / 0% CBD).
  Treatment Visit 2: Experimental: Active Alprazolam (Xanax), Placebo Cannabis Subject receives active 0.75 mg alprazolam capsule. Subject receives placebo cannabis (0% THC / 0% CBD).
  Treatment Visit 3: Experimental: Placebo Alprazolam (Xanax), Active Cannabis Subject receives alprazolam capsule containing placebo (lactose). Subject receives active cannabis (6.18% THC / <0.025% CBD).
- Sequence 2: Treatment Visit 1: Experimental: Active Alprazolam (Xanax), Placebo Cannabis Subject receives active 0.75 mg alprazolam capsule. Subject receives placebo cannabis (0% THC / 0% CBD).
  Treatment Visit 2: Experimental: Placebo Alprazolam (Xanax), Active Cannabis Subject receives alprazolam capsule containing placebo (lactose). Subject receives active cannabis (6.18% THC / <0.025% CBD).
  Treatment Visit 3: Experimental: "Sober" or Double Placebo Subject receives alprazolam capsule containing placebo (lactose). Subject receives placebo cannabis (0% THC / 0% CBD).
- Sequence 3: Treatment Visit 1: Experimental: Placebo Alprazolam (Xanax), Active Cannabis Subject receives alprazolam capsule containing placebo (lactose). Subject receives active cannabis (6.18% THC / <0.025% CBD).
  Treatment Visit 2: Experimental: "Sober" or Double Placebo Subject receives alprazolam capsule containing placebo (lactose). Subject receives placebo cannabis (0% THC / 0% CBD).
  Treatment Visit 3: Experimental: Active Alprazolam (Xanax), Placebo Cannabis Subject receives active 0.75 mg alprazolam capsule. Subject receives placebo cannabis (0% THC / 0% CBD).
- Sequence 4: Treatment Visit 1: Experimental: "Sober" or Double Placebo Subject receives alprazolam capsule containing placebo (lactose). Subject receives placebo cannabis (0% THC / 0% CBD).
  Treatment Visit 2: Experimental: Placebo Alprazolam (Xanax), Active Cannabis Subject receives alprazolam capsule containing placebo (lactose). Subject receives active cannabis (6.18% THC / <0.025% CBD).
  Treatment Visit 3: Experimental: Active Alprazolam (Xanax), Placebo Cannabis Subject receives active 0.75 mg alprazolam capsule. Subject receives placebo cannabis (0% THC / 0% CBD).
- Sequence 5: Treatment Visit 1: Experimental: Active Alprazolam (Xanax), Placebo Cannabis Subject receives active 0.75 mg alprazolam capsule. Subject receives placebo cannabis (0% THC / 0% CBD).
  Treatment Visit 2: Experimental: "Sober" or Double Placebo Subject receives alprazolam capsule containing placebo (lactose). Subject receives placebo cannabis (0% THC / 0% CBD).
  Treatment Visit 3: Experimental: Placebo Alprazolam (Xanax), Active Cannabis Subject receives alprazolam capsule containing placebo (lactose). Subject receives active cannabis (6.18% THC / <0.025% CBD).
- Sequence 6: Treatment Visit 1: Experimental: Placebo Alprazolam (Xanax), Active Cannabis Subject receives alprazolam capsule containing placebo (lactose). Subject receives active cannabis (6.18% THC / <0.025% CBD).
  Treatment Visit 2: Experimental: Active Alprazolam (Xanax), Placebo Cannabis Subject receives active 0.75 mg alprazolam capsule. Subject receives placebo cannabis (0% THC / 0% CBD).
  Treatment Visit 3: Experimental: "Sober" or Double Placebo Subject receives alprazolam capsule containing placebo (lactose). Subject receives placebo cannabis (0% THC / 0% CBD).
Period: Treatment Visit 1 (1 Day)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 2 | 2 | 1 | 1 | 1 | 1
Completed | 2 | 2 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (7 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 2 | 2 | 1 | 1 | 1 | 1
Completed | 2 | 2 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Visit 2 (1 Day)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 2 | 2 | 1 | 1 | 1 | 1
Completed | 2 | 2 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (7 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 2 | 2 | 1 | 1 | 1 | 1
Completed | 2 | 2 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Visit 3 (1 Day)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 2 | 2 | 1 | 1 | 1 | 1
Completed | 2 | 2 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects randomized completed all study arms/treatments, but in a different randomization sequence. Data was not used from subjects enrolled but not randomized.
Groups:
- Randomized Subjects: Summary of all subjects randomized. All randomized subjects completed all study arms across three treatment visits.
  "Sober" or Double Placebo: Subject received alprazolam capsule containing placebo (lactose) and 40 minutes later received placebo cannabis (0% THC / 0% CBD).
  Active Alprazolam (Xanax), Placebo Cannabis: Subject received active 0.75 mg alprazolam capsule and 40 minutes later received placebo cannabis (0% THC / 0% CBD).
  Placebo Alprazolam (Xanax), Active Cannabis: Subject received alprazolam capsule containing placebo (lactose) and 40 minutes later received active cannabis (6.18% THC / <0.025% CBD).
  Placebo (Lactose) Capsule: Single dose on two of the three visits, orally administered 40 minutes prior to cannabis dose.
  0.75 mg Alprazolam Capsule: Single dose on one of the three visits, orally administered 40 minutes prior to cannabis dose.
  Cannabis (0%/ THC / 0% CBD): Cannabis vapor was produced from 500 mg of dried plant material (0% THC / 0% CBD). Subjects inhaled using the Foltin Puff Procedure over 10 minutes. Single inflated bag/dose consumed via inhalation 40 minutes after alprazolam dose at two of the three visits.
  Cannabis (6.18% THC / <0.025% CBD): Cannabis vapor was produced from 500 mg of dried plant material (6.18% THC / <0.025% CBD). Subjects inhaled using the Foltin Puff Procedure over 10 minutes. Single inflated bag/dose consumed via inhalation 40 minutes after alprazolam dose on one of the three visits.
Arm/Group | Randomized Subjects
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Standard Deviation of Lateral Position (SDLP)
Description: The ability to keep the vehicle straight in the lane. Data is presented from the a rural drive with a concurrent divided attention task.
Time Frame: over one hour during the course of the simulator drive conducted 45 minutes post-dose at Treatment Visit 1, 2, and 3
Population: All Subjects
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | "Sober" or Double Placebo | Active Alprazolam (Xanax), Placebo Cannabis | Placebo Alprazolam (Xanax), Active Cannabis
Number analyzed (Participants) | 8 | 8 | 8
cm | 25.490 (5.737) | 37.849 (6.434) | 33.086 (12.375)

2. Secondary Outcome: Lane Exceedences
Description: Count of the number of times the simulated vehicle leaves the driving lane, will be compared across treatments. Data is from a rural drive with a concurrent divided attention task.
Time Frame: over one hour during the course of the simulator drive conducted 45 minutes post-dose at Treatment Visit 1, 2, and 3
Population: All subjects
Measure: Mean (Standard Deviation); unit: number of times vehicle departed lane
Arm/Group | "Sober" or Double Placebo | Active Alprazolam (Xanax), Placebo Cannabis | Placebo Alprazolam (Xanax), Active Cannabis
Number analyzed (Participants) | 8 | 8 | 8
number of times vehicle departed lane | 5.750 (6.251) | 36.500 (19.413) | 29.875 (48.147)

ADVERSE EVENTS:
Time Frame: Duration of study participation. Adverse Events were captured from the time of enrollment to the time of study follow-up, a maximum duration of 5 weeks.
Arm/Group | "Sober" or Double Placebo | Active Alprazolam (Xanax), Placebo Cannabis | Placebo Alprazolam (Xanax), Active Cannabis
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | "Sober" or Double Placebo (N=8) | Active Alprazolam (Xanax), Placebo Cannabis (N=8) | Placebo Alprazolam (Xanax), Active Cannabis (N=8)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs must coordinate with the government (sponsor).

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT04970342/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT04970342/ICF_001.pdf